CLINICAL TRIAL: NCT06608004
Title: Influence of Olfacto-gustatory Sensoriality on the Nutritional Status of Patients with Amyotrophic Lateral Sclerosis
Acronym: GOUSLA
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GEORGES ARSLA 2021
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient: ALS patients referred to the ALS Reference Centre at Dijon University Hospital and Lyon University Hospital
  Interventions: Other: test taking

INTERVENTIONS:
Other: test taking — Measurement of VAS for sensation of hunger, LFQP-France test, 24-hour semi-quantitative dietary recall, Assessment of energy expenditure linked to physical activity using the IPAQ (International Physical Activity Questionnaire) (only at inclusion), Screening for undernutrition risk factors using the SSQ (Social Support Questionnaire) (only at inclusion), Measurement of body composition by impedancemetry, Measurement of isometric grip strength by handgrip test, Measurement of quality of life (SF36), Study of olfacto-gustatory sensoriality (olfaction via the Sniffin' Sticks test, gustation via lingual application of impregnated strips and AHSP self-questionnaire) (carried out every other visit) and Measurement of gustatory evoked potentials in response to sugar.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease characterised by progressive diffuse muscular paralysis due to the inexorable loss of motor neurons in the primary motor cortex, the corticospinal tract, the brain stem and the spinal cord.

Over the course of the disease, when the phrenic motor neurons are involved, diaphragmatic weakness develops, leading to restrictive respiratory failure, which is the main cause of morbidity and mortality. Non-invasive ventilation (NIV) compensates for diaphragm failure and corrects the associated symptoms, and has been shown to prolong patient survival and improve quality of life.

Undernutrition is another recognised prognostic factor. Several mechanisms have been described, foremost of which are a state of hypermetabolism and a reduction in food intake secondary to chewing difficulties, dysphagia, a loss of dexterity in the upper limbs, a disturbance in salivary secretion or psychological disorders. In addition, diaphragmatic dysfunction plays a direct role in the onset of undernutrition, as compensatory contraction of the accessory neck muscles increases resting energy expenditure.

However, the hedonic sensations triggered by a meal play a role in controlling food intake beyond the simple energy balance between calorie intake and energy expenditure. Olfacto-gustatory sensoriality could therefore play a role in the nutritional status of patients suffering from ALS.

Diaphragmatic dysfunction may also influence nutritional status by other mechanisms. For example, the reduction in inspiratory capacity associated with diaphragmatic insufficiency reduces olfaction in a group of tetraplegic patients. Central sensory impairment could exacerbate this phenomenon. Although it is conventionally considered that there are no sensory manifestations during the course of ALS, minor but diffuse abnormalities of the nerves and sensory action potentials have been observed. A central alteration in olfacto-gustatory sensoriality could be part of the neurological manifestations of ALS. In addition, olfactory deficits occur in other neuromuscular diseases with central involvement, such as myasthenia, Parkinson's or Alzheimer's disease, in the absence of concomitant cognitive or diaphragmatic impairment.

Our hypothesis is that impaired olfacto-gustatory function favours the onset of undernutrition in ALS.

Current nutritional management consists of ensuring adequate calorie intake by prescribing oral food supplements or inserting a gastrostomy. Taking personalised account of food preferences during dietary advice or of a potential olfacto-gustatory deficit, by reinforcing smells or tastes during food consumption, would be an interesting additional therapeutic avenue for improving patients' nutritional status, quality of life and prognosis

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria*:

* Incident cases of definite or probable ALS according to El-Escorial criteria (3) followed up at the participating regional centre of competence
* Patient aged over 18
* Patient fluent in French
* Patient having given oral consent

Exclusion Criteria:

* Patients with an acute infection undergoing antibiotic treatment at the time of inclusion
* Patients with psychiatric, cognitive or neurological disorders making it impossible to assess food preferences
* Patient with a known food allergy
* Patients with excessive alcohol consumption (≥ 10 standard drinks per week)
* Patients who have stopped smoking for less than 1 month
* Patients with severe bulbar involvement from the outset, preventing swallowing, patients with aphagia or patients eating exclusively via a gastrostomy
* Patient with severe diaphragmatic impairment requiring NIV from the outset
* Person not affiliated to or not benefiting from a social security scheme
* Person under legal protection (curatorship, guardianship)
* Persons subject to a legal protection measure
* Pregnant women, women in labour or breastfeeding mothers
* An adult who is incapable or unable to give consent
* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALS will be referred to the regional reference centre for treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The measurement of implicit wanting | Through study completion, on average of 12 months
  It is calculated for each food category (sweet-poor-fat, sweet-rich-fat, salty-poor-fat and salty-rich-fat) using the Leeds Food Preference Questionnaire (LFQP-France), which measures food preferences. This is a standardised computerised test (32), adapted to French cultural habits. It consists of presenting patients with photos of foods rich in carbohydrates, proteins or lipids.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France